CLINICAL TRIAL: NCT05358847
Title: Safety and Efficacy of Sofwave Treatment for Improvement of Cellulite Appearance
Brief Title: Treatment for Cellulite Appearance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sofwave Medical LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sofwave08
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-04

CONDITIONS: Cellulite
Keywords: upper thigh, buttock, skin laxity
MeSH Terms: conditions — Cellulite; Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cellulite (Experimental)
  Interventions: Device: Sofwave

INTERVENTIONS:
Device: Sofwave — The Sofwave System, comprised of an applicator and a console, generates high intensity, non-focused ultrasonic energy which can be delivered percutaneously to tissues.
  Other Names: SUPERB

SUMMARY:
Open-label, non-randomized, prospective, multi-center, self-controlled clinical study with masked evaluation.

DETAILED DESCRIPTION:
Eligible patients will receive 2 treatments (4-6 weeks apart) on one side (right or left) of the lateral/ posterior upper thigh / buttocks using Sofwave System.

Treatment may be administered after the enrollment and screening at the first visit, or it may occur later following the enrollment and screening activities based on site scheduling availabilities.

All patients will return to the clinic for one follow up visits at 3 months ± 3 weeks post last treatment (FU1). Optionally, additional follow-up visit will be conducted 6 (± 4 weeks) months following end of treatment (FU2).

Methodology described in the protocol to evaluate efficacy and safety of treatments will be carried out at each visit at the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects > 18 years of age and < 60 years of age
2. Not pregnant or lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide) or abstinence.
3. Have visible cellulite in the upper thigh and/or buttock areas.
4. Seeking treatment of cellulite in the upper thigh and/or buttock areas.
5. Stable weight nominally ±5% for at least past 6 months
6. Subject agrees to maintain her weight (i.e., within 5% of total body weight) by not making any major changes in their diet or exercise routine during the study course.
7. Subject did not undergo invasive or energy-based cellulite treatments (liposuction, subcision, RF, laser, ESWT, etc.) for the prior 12 months.
8. Subject did not use topical based cellulite treatments for prior 6 months and will not use during the trial (except for the study related procedures)
9. Subject agrees not to undergo any other cellulite treatments for a period of 6 months following Sofwave treatment
10. Willing to have photographs of the treated areas. Agree for de-identified study images to be used in evaluations, publications, and presentations.
11. Able and willing to comply with all visits, treatments and evaluations schedules and requirements.
12. Able to understand and provide written Informed Consent.

Exclusion Criteria:

1. Pregnant or planning to become pregnant during the duration of the study, having given birth less than 3 months ago, and/or breast feeding
2. Currently heavy smoker or has history of heavy smoking (25 cigarettes per day or more) in past 10 years
3. BMI>=30kg/m2
4. Non-stable weight nominally ±5% for at least past 6 months
5. Currently taking or has taken diet pills or weight control supplements within the past month
6. History of severe migraine tendency
7. History of Epileptic seizures
8. History of chronic drug or alcohol abuse
9. History of coagulopathy(ies) and/or on anticoagulant medication
10. History of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising
11. Medical disorder that would hinder the wound healing or immune response (such as blood disorder, inflammatory disease, etc.)
12. Active implanted device such as a pacemaker, defibrillator, cochlear implants, nerve/brain stimulators or drug delivery system
13. Known allergy to lidocaine or epinephrine or antibiotics
14. Active malignancy or history of malignancy in the past 5 years
15. Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), lupus, porphyria, or pertinent neurological disorders (i.e. any disease state that in the opinion of the investigator may interfere with the anesthesia, treatment, or healing process)
16. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications
17. Suffering from hormonal imbalance, whether related to thyroid, pituitary, or androgen
18. History of significant lymphatic drainage problems
19. History of epidermal or dermal disorders (particularly involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders.
20. Skin disorders (skin infections or rashes, extensive scarring, psoriasis, etc.) in the treatment area.
21. Severe solar elastosis on the intended to treat area.
22. Significant scarring, atrophic scars in the area to be treated, or has a history of atrophic scars or keloids or prone to bruising
23. Tattoo or former tattoo at or near treatment area
24. Presence of an implant (metal or plastic) in or adjacent to area of intended treatment (vascular stent, or implants in the hips, knees, etc)
25. Inability to understand the protocol or to give informed consent
26. On-going use of psychiatric medication
27. Unable or unwilling to comply with the study requirements and procedures
28. Unwilling to have research photos taken of treatment areas
29. Currently enrolled in a clinical study of any other unapproved investigational drug or device
30. Any other condition that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Rate of improvement in the appearance of cellulite on the upper thigh/buttock area | 3 months post treatment follow-up visit.
  following Sofwave treatments based on 6 points simplified Cellulite Severity Scale (CSS), as evaluated by independent masked reviewers.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Laser & Skin Surgery Center of Northern California, Sacramento, California
  - UnionDerm, New York, New York
  - Laser & Skin Surgery Center of New York®, New York, New York
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided